CLINICAL TRIAL: NCT00371163
Title: Molecular and Cellular Characterization of Spongiotic Dermatitis
Acronym: Spongiotic
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 200614530
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Atopic Dermatitis; Psoriasis; Contact Dermatitis
Keywords: Identification of genes by microarray analyses.
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis; Dermatitis, Contact

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Contact Dermatitis: Males or females with contact dermatitis
- Psoriasis: Males or females with psoriasis
- No skin disease: Males or females with no skin diseases
- Atopic Dermatitis: Males of females with atopic dermatitis

SUMMARY:
Spongiotic dermatitis is the histopathologic diagnosis commonly issued by dermatopathologists that encompasses atopic dermatitis, contact dermatitis, and other forms of eczematous dermatitis.

The information obtained will assist in development of diagnostic methods for differentiation of the types of spongiotic dermatitis. This study also has the potential to lead to the dissection of pathologic pathways involved in these diseases and development of novel therapeutic agents.

DETAILED DESCRIPTION:
Spongiotic dermatitis is the histopathologic diagnosis commonly issued by dermatopathologists that encompasses atopic dermatitis, contact dermatitis, and other forms of eczematous dermatitis. Atopic dermatitis is a chronic, relapsing inflammatory disease characterized by pruritic, scaly, red, eczematous skin lesions, and a personal or family history of atopy. Patients affected by atopic dermatitis experience significant morbidity from extreme pruritus, recurrent cutaneous infections, and extensive and/or disfiguring skin lesions. Allergic contact dermatitis typically manifests as pruritus and vesicular or eczematous lesions associated with direct exposure to environmental haptenic allergens.

The specific aims of this research are:

1. Identification of genes differentially expressed in atopic dermatitis, contact dermatitis, and psoriasis by microarray analyses.
2. Confirmation of protein expression profiles in atopic and contact dermatitis, and psoriasis by immunohistochemical analyses.
3. Identification of disease-specific potential diagnostic markers in plasma and PBMC.

The information obtained will assist in development of diagnostic methods for differentiation of the types of spongiotic dermatitis. This study also has the potential to lead to the dissection of pathologic pathways involved in these diseases and development of novel therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Atopic Dermatitis: Subjects will be identified based on the Hanifin criteria of atopic dermatitis. Subjects will be adults with a history of atopic dermatitis since childhood, who continue to have symptoms and signs of atopic dermatitis. They must have active lesions and should not be on systemic therapy.
2. Contact Dermatitis: Subjects will be adults with history of contact dermatitis to common allergens. They will undergo patch testing to common allergens and the sites of positive reactions will be considered as lesional skin.
3. Psoriasis: Subjects will be adults with chronic disease, who have active skin lesions with a characteristic morphology.

Subjects will be asked to discontinue topical medications at least to parts of the skin where biopsies will be taken, one week prior to biopsy.

-

Exclusion Criteria:

* Patients on systemic treatment of their skin diseases within the past one month.
* A history of significant neurologic, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic diseases.
* Abnormal hepatic function or renal function (creatinine or BUN is > 1.2 times the upper level of the normal range for the laboratory where the testing is done).
* Abnormal blood counts (WBC < 4 x 103/mm3; platelet < 100 x 103/mm3; hemoglobin < 11g/dl).
* History of alcohol or drug abuse.
* Known hepatitis or HIV.
* Pregnant women (as determined by serum pregnancy test).
* Significant allergic or adverse reaction to local anesthetics.
* Blood clotting disorder.
* Faintness or vasovagal reaction with blood draws or procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Males or females aged 18-55 with either contact dermatitis, psoriasis, atopic dermatitis, or no skin disease.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2006-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Identification of disease-specific potential diagnostic markers in plasma and PBMC. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tong Liu, M.D., Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical